CLINICAL TRIAL: NCT06828822
Title: CIRCLE : CongenItal Naevus Cohort for Longitudinal Evaluation
Brief Title: CongenItal Naevus Cohort for Longitudinal Evaluation
Acronym: CIRCLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RC24_0532
Record Dates: First submitted 2025-01-29; First posted 2025-02-14 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Naevi; Neurodevelopmental Disorder; Congenital Nevus
Keywords: Congenital Nevus; Neurodevelopmental Disorder
MeSH Terms: conditions — Nevus; Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child with a congenital nevus (Experimental)
  Interventions: Other: Neurodevelopmental assessment; Other: Patient quality of life assessment
- Legal representatives (Other)
  Interventions: Other: Meeting with the parents

INTERVENTIONS:
Other: Neurodevelopmental assessment — This assessment will be conducted using the ASQ-3 test. (ASQ-3 stands for Ages and Stages Questionnaires, Third Edition, which is a common screening tool for evaluating developmental progress in young children.)
  Arms: Child with a congenital nevus
Other: Meeting with the parents — This meeting will evaluate the parents' acceptance of the lesion and their quality of life using the MARKS test (Measure of Acceptance of Skin Marks). The results will provide insights into how the parents perceive the lesion and how it impacts their daily lives.
  Arms: Legal representatives
Other: Patient quality of life assessment — Collection of patient quality of life data
  Arms: Child with a congenital nevus

SUMMARY:
Congenital Nevus (CN) is a pigmented skin lesion present at birth, which grows in size as the child grows. It can vary in appearance and is classified by its size, from small (less than 1.5 cm) to giant (greater than 40 cm). CN is associated with genetic mutations, mainly in the NRAS/BRAF genes.

A large CN can lead to several clinical issues, including:

Risk of neurological disorders: Large CN can be associated with neurological abnormalities such as neuro-meningeal melanosis, hydrocephalus, or brain malformations. These conditions may cause early neuro-developmental delays. The risk is not well understood and requires further studies.

Risk of melanoma: The risk of developing melanoma is higher for a large CN but remains low for smaller ones. Increased monitoring is necessary during the early years for large and giant CN.

Psycho-social impact: Parents often experience significant anxiety at birth due to the cancer risk and social stigma. As the child grows, a visible CN may impact their quality of life, particularly socially at school.

Management of CN remains controversial, especially for those of medium to giant size or with multiple satellites. There is an urgent need for further research to clarify best practices in monitoring and treatment, including the need for routine brain imaging and criteria for surgical intervention.

Ultimately, this study aims to deepen our understanding of CN, its associated neurological and melanoma risks, and the psycho-social challenges it poses, while striving to establish clear, evidence-based guidelines for monitoring and treatment to enhance patient outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient under 2 years old.
* Patient with a medium, large, or giant congenital nevus (CN) according to the Krengel classification, either single or multiple.
* Patient affiliated with social security.
* Patient whose legal representatives consent to their child's participation in the project.

Exclusion Criteria:

* Patient with light brown spots or pigmented lesions not classified as nevi.
* Patient for whom It is impossible to establish annual follow-up.
* Patient whose parents do not speak French.

Ages: 0 Years to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 819 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2031-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Determine the prevalence of neurodevelopmental abnormalities in infants and young children with medium to giant congenital nevus, and according to nevus characteristics (size, number), at the age of 3 years. | 3 years.
  This assessment will be conducted using the ASQ-3 (Ages and Stages Questionnaires, Third Edition).

SECONDARY OUTCOMES:
The occurrence of other neurological abnormalities (early epilepsy, etc.), screening for psychomotor developmental delays. | 3 years
The prevalence of neurological abnormalities on MRI (Magnetic Resonance Imaging), both absolutely and according to the characteristics of the congenital nevus. | 3 years.
The occurrence of early melanoma or another tumor. | 3 years.
The evolution of the clinical characteristics of the congenital nevus (size, color, texture, number of satellites), and associated functional signs (pruritus). | 3 years.
  According to the Krengel classification 1 (size, projected adult size, number of satellites) and assessment of color, roughness, hair growth, pruritus/eczematization, and proliferative nodules.
Description of the histopathological characteristics of the congenital nevus (if available) following excision or biopsy. | 3 years.
  If an excision or biopsy is performed, it will be possible to provide the histopathological characteristics of the congenital nevus (CN).
Description of the molecular characteristics of the congenital nevus (if available) following excision or biopsy. | 3 years.
  If an excision or biopsy is performed, it will be possible to provide the molecular characteristics of the congenital nevus (CN).
Parental satisfaction of cares management and surgery. | 3 years.
  Parental satisfaction with the management and surgery, if performed, and evaluation of the patient's satisfaction with the intervention using a Visual Analog Scale (VAS).
Lesion acceptance and quality of life. | 3 years.
  The parents' acceptance of the lesion and their quality of life will be evaluated using the MARKS test (Measure of Acceptance of Skin Marks). The results will provide insights into how the parents perceive the lesion and how it impacts their daily lives.
Identification of factors influencing the clinical care pathway and their correlation on health outcomes. | 3 years.
Identification of the patient's well-being using the Cartoon CDLQI test. | 3 years.
  The Cartoon Children's Dermatology Life Quality Index (Cartoon CDLQI) is a version of the Children's Dermatology Life Quality Index (CDLQI) designed to make assessing the quality of life in children with skin diseases more engaging and accessible for younger children. (Scale from 1 to 4 ; with 4 being the worst outcome ( "a lot" ) and 1 being the best ("not at all").

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Grasse Hospital, Nice, Alpes-Maritimes
  - Nice University Hospital and Lenval Hospital, Nice, Alpes-Maritimes
  - Marseille University Hospital, Marseille, Bouches-du-Rhône
  - Dijon University Hospital, Dijon, Côte-d'Or
  - La Réunion University Hospital, La Réunion, Département Et Région D'outre-mer
  - Brest University Hospital, Brest, Finistère
  - Bordeaux University Hospital, Bordeaux, Gironde
  - Toulouse University Hospital, Toulouse, Haute-Garonne
  - Rennes University Hospital, Rennes, Ille-et-Vilaine
  - Tours University Hospital, Tours, Indre-et-Loire
  - Nantes University Hospital, Nantes, Loire Atlantique
  - Angers University Hospital, Angers, Maine et Loire
  - Nancy University Hospital, Nancy, Meurthe-et-Moselle
  - Saint Vincent de Paul Hospital, Lille, Nord
  - Paris Necker Hospital, Paris, Paris

IPD SHARING:
Plan to Share IPD: Undecided